CLINICAL TRIAL: NCT01370408
Title: A Unique Schedule of Palonosetron, Ondansetron, and Dexamethasone for the Prevention of Delayed Nausea and Vomiting in Patients Receiving Moderately Emetogenic Myeloablative Chemotherapy
Brief Title: Palonosetron, Ondansetron, and Dexamethasone for Delayed Nausea and Vomiting in Autologous Transplant Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northside Hospital, Inc. (Other)
Collaborators: Blood and Marrow Transplant Group of Georgia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NSH 940
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: Autologous stem cell transplant; BEAM; Oral busulfan; Cyclophosphamide; Etoposide; Carboplatin; melphalan
MeSH Terms: conditions — Vomiting | interventions — Palonosetron; Ondansetron; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Palonosetron (Experimental): All patients will receive the following medications prior to and during their high dose chemotherapy for autologous stem cell transplantation
  Prior to IV chemotherapy - ondansetron 8mg IV & Dexamethasone 10 mg IV on the last day of chemotherapy - Palonosetron .25 mg IV, dexamethasone 10mg IV Day 1-2 after IV chemotherapy - Dexamethasone 8 mg PO
  Interventions: Drug: Palonosetron; Drug: ondansetron; Drug: Dexamethasone

INTERVENTIONS:
Drug: Palonosetron — Prior to IV chemotherapy - ondansetron 8mg IV & Dexamethasone 10 mg IV On the last day of chemotherapy - Palonosetron .25 mg IV, dexamethasone 10mg IV Day 1-2 after IV chemotherapy - Dexamethasone 8 mg PO
  Other Names: Aloxi
Drug: ondansetron — Prior to IV chemotherapy - ondansetron 8mg IV & Dexamethasone 10 mg IV On the last day of chemotherapy - Palonosetron .25 mg IV, dexamethasone 10mg IV
  Other Names: zofran
Drug: Dexamethasone — Prior to IV chemotherapy - ondansetron 8mg IV & Dexamethasone 10 mg IV On the last day of chemotherapy - Palonosetron .25 mg IV, dexamethasone 10mg IV
  Other Names: Dex

SUMMARY:
In this study, patients will receive ondansetron 8mg and dexamethasone 10mg intravenously 30 minutes prior to myeloablative preparative chemotherapy until the last day of chemotherapy. On the final day of chemotherapy, palonosetron 0.25mg and dexamethasone 10mg will be administered intravenously 30 minutes prior to the chemotherapy. If the chemotherapy regimen is only 1 day of the chemotherapy then only palonosetron and dexamethasone will be administered 30 minutes prior to chemotherapy. Dexamethasone 8mg once daily will be given orally for 2 days following chemotherapy.

DETAILED DESCRIPTION:
In order to decrease this delayed CINV, the investigators have developed a unique schedule of antiemetics that takes advantage of palonosetron's long elimination half-life (40 hours). In this study, patients will receive ondansetron 8mg and dexamethasone 10mg intravenously 30 minutes prior to myeloablative preparative chemotherapy until the last day of chemotherapy. On the final day of chemotherapy, palonosetron 0.25mg and dexamethasone 10mg will be administered intravenously 30 minutes prior to the chemotherapy. If the chemotherapy regimen is only 1 day of the chemotherapy then only palonosetron and dexamethasone will be administered 30 minutes prior to chemotherapy. Dexamethasone 8mg once daily will be given orally for 2 days following chemotherapy. The investigators hypothesize that this antiemetic schedule will significantly reduce the delayed CINV compared to historical controls

ELIGIBILITY:
Inclusion Criteria:

* candidate for high-dose chemotherapy and autologous hematopoietic stem cell transplantation
* Karnofsky performance status >/= 60%
* scheduled to receive one of the following conditioning regimens
* BEAM
* Oral Busulfan/cyclophosphamide with or without etoposide
* Carboplatin/Etoposide
* Melphalan
* Negative pregnancy test
* Must be able to complete a daily nausea/vomiting questionnaire and Quality of Life

Exclusion Criteria:

* Active infection requiring IV antibiotics
* Known active hepatitis B and/or hepatitis C or HIV infection
* prior non-hematological malignancies at other sites except surgically treated non-melanoma skin cancer, superficial cervical cancer or other cancer from which the patient had been disease free for >/= 5 years
* Uncontrolled medical problems including any of the following
* Diabetes mellitus
* Cardiac, pulmonary, hepatic or renal disease
* myocardial infarction within the past 6 months
* Morbid obesity (BMT >40)
* History of CNS metastases, psychiatric or CNS disorders interfering with the ability to comply with the study
* Known hypersensitivity to 5-HT3 antagonists, dexamethasone and/or their components
* Intrathecal therapy within 24 hours before starting preparative regimen
* Receiving any antiemetic therapy 24 hours before starting preparative regimen
* Any 5-HT3 antagonist used as a rescue medication

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2012-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott R Solomon, MD, Principal Investigator — Blood and Marrow Transplant Group of Georgia
Locations (1):
- Northside Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Palonosetron: All patients will receive the following medications prior to and during their high dose chemotherapy for autologous stem cell transplantation
  Day x-y of IV chemotherapy - ondansetron 8mg IV & Dexamethasone 10 mg IV Day z (last day of chemotherapy) - Palonosetron .25 mg IV, dexamethasone 10mg IV Day 1-2 after IV chemotherapy - Dexamethasone 8 mg PO
  Palonosetron, ondansetron, dexamethasone: Day x-y of IV chemotherapy - ondansetron 8mg IV & Dexamethasone 10 mg IV Day z (last day of chemotherapy) - Palonosetron .25 mg IV, dexamethasone 10mg IV Day 1-2 after IV chemotherapy - Dexamethasone 8 mg PO
Period: Overall Study
Arm/Group | Palonosetron
Started | 85
Completed | 76
Not Completed | 9
Not completed — treatment failure | 9

BASELINE CHARACTERISTICS:
Arm/Group | Palonosetron
Number analyzed (Participants) | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 56
  >=65 years | 29
Age, Continuous [Median (Full Range); unit: years] | 57 [20 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 47
Region of Enrollment [Number; unit: participants]
  United States | 85

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate for Delayed Chemotherapy Induced Nausea & Vomiting
Description: Proportion of patients achieving a delayed CINV complete response (CR) defined as no emetic episode and no use of rescue medications during the 24-120 hour period post chemotherapy.
Time Frame: 120 hours
Measure: Number; unit: participants
Arm/Group | Palonosetron
Number analyzed (Participants) | 85
participants | 13

2. Secondary Outcome: Complete Remission During Acute Phase Post-chemotherapy
Description: Proportion of patients achieving an acute CINV CR during the acute phase post -chemotherapy (0-24 hours)
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Palonosetron
Number analyzed (Participants) | 85
participants | 33

3. Secondary Outcome: Complete Remission During Overall Chemotherapy Time Period
Description: Proportion of patients achieving a CR during the cumulative overall 0-120 hour time period
Time Frame: 120 hours
Measure: Number; unit: participants
Arm/Group | Palonosetron
Number analyzed (Participants) | 85
participants | 10

4. Secondary Outcome: Complete Control Rate for Nausea & Vomiting
Description: Complete control rate (CC; defined as no emetic episodes, no rescue medication use, and no more than mild nausea)
Time Frame: 120 hours
Measure: Number; unit: participants
Arm/Group | Palonosetron
Number analyzed (Participants) | 85
participants | 8

5. Secondary Outcome: Emetic Episodes
Description: Number of emetic episodes
Time Frame: 120 Hours
Measure: Mean (Full Range); unit: episodes
Arm/Group | Palonosetron
Number analyzed (Participants) | 85
episodes | 1.7 [1 to 24]

6. Secondary Outcome: Patients Who Experience First Emetic Episode Within 24 Hours
Description: Number of patients with first emetic episode experienced within 24 hours
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Palonosetron
Number analyzed (Participants) | 85
participants | 15

7. Secondary Outcome: Number of Patients That Required First Administration of Rescue Medication Within 24 Hours
Description: Number of patients who required the use of rescue medication (lorazepam, prochlorperazine, promethazine, metoclopramide, scopolamine, or dronabinol) within the first 24 hours
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Palonosetron
Number analyzed (Participants) | 85
participants | 46

8. Secondary Outcome: Number of Patients That Experience Treatment Failure Within the First 24 Hours
Description: Number of patients with first emetic episode or time to administration of rescue therapy, whichever occurred first, within the first 24 hours
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Palonosetron
Number analyzed (Participants) | 85
participants | 49

ADVERSE EVENTS:
Arm/Group | Palonosetron
Serious Adverse Events (participants affected / at risk) | 0/85
Other Adverse Events (participants affected / at risk) | 85/85
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Palonosetron (N=85)
abdominal distension (Gastrointestinal disorders) | 6
abdominal cramping (Gastrointestinal disorders) | 19
increased alkaline phosphatase (Hepatobiliary disorders) | 11
increased ALT (Hepatobiliary disorders) | 8
neutropenia (Blood and lymphatic system disorders) | 65
anemia (Blood and lymphatic system disorders) | 53
anorexia (Gastrointestinal disorders) | 15
anxiety (Psychiatric disorders) | 32
increased AST (Hepatobiliary disorders) | 19
abdominal tenderness (Gastrointestinal disorders) | 7
back pain (Musculoskeletal and connective tissue disorders) | 5
rectal bleeding (Gastrointestinal disorders) | 6
bruising (Skin and subcutaneous tissue disorders) | 5
chills (Investigations) | 10
constipation (Gastrointestinal disorders) | 18
cough (Respiratory, thoracic and mediastinal disorders) | 8
decreased appetite (Gastrointestinal disorders) | 37
deconditioning (Investigations) | 5
diarrhea (Gastrointestinal disorders) | 48
dizziness (Nervous system disorders) | 20
dry skin (Skin and subcutaneous tissue disorders) | 5
dry mouth (Gastrointestinal disorders) | 15
dysuria (Renal and urinary disorders) | 11
lower extremity edema (Cardiac disorders) | 15
fatigue (Investigations) | 56
gastroesophageal reflux disease (Gastrointestinal disorders) | 11
headache (Nervous system disorders) | 24
hiccups (Gastrointestinal disorders) | 7
hyperbilirubinemia (Hepatobiliary disorders) | 14
hyperglycemia (Metabolism and nutrition disorders) | 47
hypermagnesemia (Metabolism and nutrition disorders) | 8
hypernatremia (Metabolism and nutrition disorders) | 11
hypertension (Cardiac disorders) | 9
hypoalbuminemia (Hepatobiliary disorders) | 33
hypocalcemia (Metabolism and nutrition disorders) | 33
hypoglycemia (Metabolism and nutrition disorders) | 6
hypokalemia (Metabolism and nutrition disorders) | 23
hypomagnesemia (Metabolism and nutrition disorders) | 9
hyponatremia (Metabolism and nutrition disorders) | 14
hypotension (Cardiac disorders) | 12
insomnia (Psychiatric disorders) | 23
lymphopenia (Blood and lymphatic system disorders) | 24
memory changes (Nervous system disorders) | 6
mouth pain (Gastrointestinal disorders) | 11
mouth sores (Gastrointestinal disorders) | 9
mucositis (Gastrointestinal disorders) | 19
nausea (Gastrointestinal disorders) | 74
neutropenic fever (Infections and infestations) | 14
peripheral neuropathy (Nervous system disorders) | 7
pruritus (Skin and subcutaneous tissue disorders) | 6
rash (Skin and subcutaneous tissue disorders) | 15
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 5
shortness of breath with exertion (Respiratory, thoracic and mediastinal disorders) | 12
sore throat (Gastrointestinal disorders) | 17
tachycardia (Cardiac disorders) | 19
taste alteration (Gastrointestinal disorders) | 5
throat pain (Gastrointestinal disorders) | 8
thrombocytopenia (Blood and lymphatic system disorders) | 53
urinary frequency (Renal and urinary disorders) | 7
vomiting (Gastrointestinal disorders) | 49
leukopenia (Blood and lymphatic system disorders) | 74
generalized weakness (Investigations) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No